## **Informed Consent for Nurses**

Title: A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses

NCT Number: Not Available as yet

Document Date
December 5, 2025

# **GENERAL CONSENT FOR PARTICIPATION IN RESEARCH** موافقة عامة بالمشاركة في بحث

Title of Research: A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses

عنوان البحث: تجربة سريرية عشوانية مضبوطة حول تطبيق الذكاء الاصطناعي في تقييم الجلد للوقاية من تقرحات الفراش وتحديد مراحلها بواسطة ممرضي وحدات العناية المركزة

Part I - Research Participant Information Sheet:

الجزء الأول - معلومات للمشارك في البحث:

أنت مدعو للمشاركة في بحث علمي

You are invited to participate in a Scientific research project

A. Purpose of the Research: is to examine the effectiveness and impact of AI-assisted skin assessments and PI staging in critical care settings, by comparing its accuracy, reliability, and nurses' confidence and knowledge with those of traditional assessment methods employed by critical care nurses.

أ. الغرض من البحث: تهدف هذه الدراسة إلى تقييم فعالية وتأثير التقييمات الجلدية المدعومة بالذكاء الاصطناعي وتحديد مراحل تقرحات الفراش في وحدات العناية المركزة، من خلال مقارنة دقتها وموثوقيتها وثقة الممرضين ومعرفتهم بها مع طرق التقييم التقليدية التي يستخدمها ممرضو العناية المركزة

B. Description of the Research:

As part of this study, you will be randomly assigned to one of two groups. One group, called the control group, will undergo skin assessments conducted solely by the nurse using the standard approach. The other group, called the intervention group, will have nurses who use an Artificial Intelligence (AI) device, which involves taking a photograph of the patient's skin and applying the Al tool to assist in the assessment. In both groups, a Wound Care Specialist will review the assessments to ensure that the most accurate findings are used when developing the treatment plan.

Before the intervention begins, participants in both groups will complete a short questionnaire to measure their knowledge of and confidence in performing skin assessments. Following this, all participants will receive training provided by the Wound Care Department on skin assessment and pressure injury staging. Nurses in the intervention group will receive additional training on how to use the AI tool effectively. After the intervention, the questionnaire on knowledge and confidence in skin assessment will be repeated to assess any improvements.

ب. وصف البحث:

كجزء من هذه الدراسة، سيتم توزيعك عشوانيًا إلى إحدى مجموعتين. المجموعة الأولى، وتسمى مجموعة الضبط، سيُجرى فيها تقييم الجلد من قبل الممرضة فقط باستخدام الطريقة المعتادة. أما المجموعة الثانية، وتسمى مجموعة التدخل، فسيقوم فيها الممرضون باستخدام جهاز الذكاء الاصطناعي، والذي يتضمن التقاط صورة لجلد المريض وتطبيق أداة الذكاء الاصلطناعي للمساعدة في التقييم. في كلتا المجموعتين، سيقوم أخصاني العناية بالجروح بمرّاجعة التقييمات الَّتأكد من اسّتخدام

أدق النتائج عند وضع خطة العلاج. قبل بدء التدخل، سيطلب من المشاركين في كلتا المجموعتين تعبئة استبيان قصير لقياس معرفتهم وتقتهم في أداء تقييمات الجلد بعد ذلك، سيحصل جميع المشاركين على تدريب مقدم من قسم العناية بالجروح حول تقييم الجلد وتصنيف مراحل إصابات تقرحات الفراش. وسيحصل الممرضون في مجموعة التدخل على تدريب إضافي حول كيفية استخدام أداة الذكاء الاصطناعي بفعالية. بعد انتهاء التدخل، سيتم إعادة الاستبيان المتعلق بالمعرفة والثقة في تقييم الجلد لقياس أي تحسن تحقق.

#### C. Potential Benefits:

Participation in this study may contribute to the prevention of pressure injuries by improving the accuracy of skin assessments and enhancing nurses' knowledge and confidence in assessment practices. While individual participants may not directly benefit, the ج. الفوائد المحتملة:

قد تساهم المشاركة في هذه الدراسة في الوقاية من إصابات تقرحات الفراش من خلال تحسين دقة تقييمات الجلد وتعزيز معرفة الممرضين وثقتهم في ممارسات التقييم. وعلى الرغم من أن المشاركين الأفراد قد لا يستفيدون بشكل مباشر، إلا أن نتائج الدراسة قد تسهم في تحسين نتائج المرضى ودعم دمج الأدوات المبتكرة في الممارسة

This Informed Consent Form (ICF) is approved by the KFSHRC -IRB

ICF Version No.: 1.0

IRB # 2251201

Approval Dated

From: 27 October 2025

To: 31 August 2026



INFORMED CONSENT FOR RESEARCH (Cross out the nonapplicable)\*

إذن ناف للجهالة بالموافقة على بحث (اشطب ما لا ينطبق) \*

findings have the potential to improve patient outcomes and support the integration of innovative tools in clinical practice.

#### D. Potential Risks and Discomforts:

The study poses no physical risks. However, some participants may feel uneasy when answering the knowledge and confidence questionnaire, as it could be perceived as an evaluation of their professional competence. To minimize this, responses will be anonymous and used solely for research purposes. Results will not be shared with Nurse Managers or used in staff performance evaluations.

## E. Voluntary Participation:

Participation in this study is voluntary. You will not suffer penalty nor loss of any benefits to which you are entitled for, if you decide not to participate.

Significant new findings developed during the course of the study, which might be expected to affect your willingness to continue to participate in the study, will be provided to you.

A signed copy of consent form will be given to you.

#### F. Alternative to Participation (if applicable):

Withdrawal from or not participating in this research study will not affect your ability to obtain alternative methods of medical care available at King Faisal and Research Centre (General Organization) - Jeddah

#### G. Termination of Participation (where applicable):

Taking part in this study is completely voluntary. You have the right to stop participating at any time, for any reason, and this will not affect your employment at the hospital.

#### د. المخاطر والانزعاجات المحتملة:

لا تشكل الدر اسة أي مخاطر جسدية. ومع ذلك، قد يشعر بعض المشاركين بعدم الارتياح عند الإجابة على استبيان المعرفة والثقة، إذ قد يُنظر إليه على أنه تقييم لكفاءتهم المهنية. وللتقليل من ذلك، ستكون الإجابات مجهولة الهوية وستُستخدم لأغراض البحث فقط. ولن يتم مشاركة النتائج مع مديري التمريض أو استخدامها في تقييم أداء المو ظفين.

#### ه. المشاركة الطوعية:

المشاركة في هذه الدراسة طوعية. ولن تتعرض لأي عقوبة أو فقدان لأي من المزايا التي يحق لك الحصول عليها إذا قررت عدم المشاركة.

سيتم إبلاغك بأي نتانج جديدة وهامة يتم التوصل إليها أثناء سير الدراسة، والتي قد تؤثر على رغبتك في الاستمرار بالمشاركة فيها.

سيتم تزويدك بنسخة موقعة من هذا الإقرار

و. البدائل عن المشاركة (إن وجد):

إن قرارك بعدم الإشتراك أو بالإنسحاب من الدراسة لن يؤثر على تلقيك لخدمات علاجية بديلة متوفرة في مستشفى الملك فيصل التخصصي و مركز الابحاث بجدة (مؤسسة عامة).

#### ز. إنهاء المشاركة (عند الضرورة):

المشاركة في هذه الدراسة طوعية تمامًا. ليك الحق في التوقيف عن المساركة في أي وقت ولأي سبب، ولن يوثر ذلك على وظيفتك في

This Informed Consent Form (ICF) is approved by the KFSHRC -IRB

ICF Version No.: 1.0

IRB # 2251201

Approval Dated:

From: 27 October 2025

To: 31 August 2026 5



## H. Confidentiality:

Your identity as a participant in this research study, will remain confidential with respect to any publications of the results of this study. However, your identity may be reviewed by the principal investigator/ delegate involved in this research, the Research Ethics Committee, or the agency sponsoring this research in accordance with applicable laws and regulations.

#### I. Compensation/ Treatment:

Financial compensation from KFSHRC-J, however, is not available.

#### J. Cost/s Reimbursements:

You will not be not be expected to pay any fees related to your participation in this study.

# K. Contact Person(s):

For any specific questions regarding this study or in the event of a research-related injury, please contact the pricipal investigator/delegate, , Dr Jennifer de Beer phone No. 012667-7777 Ext. 66403

For general questions concerning research at KFSHRC-Jeddah, you may call the research coordinator telephone # 012667-7777

Ext...63537. or the Research Ethics Committee telephone# 966114424528

#### ح. السرية:

ستظل هويتك كمشارك في هذه الدراسة البحثية سرية فيما يتعلق بأي منشورات لنتائج هذه الدراسة. ومع ذلك، قد يتم الاطلاع على هويتك من قبل الباحث الرنيسي أو من يفوضه، أو من قبل لجنة أخلاقيات البحث، أو الجهة الراعية لهذه الدراسة، ونلك وفقًا للأنظمة والقوانين المعمول بها

ط. التعويضات/ العلاج:

لن يتم توفير تعويض مالي من مستشفى الملك فيصل التخصصى ومركز الأبحاث - جدة.

ي التكاليف/ التعويض المالي:

لنَّ يُطلب منك دفع أي رسوم تتعلق بمشاركتك في هذه الدراسة.

# ك الأشخاص الذين يمكن الاتصال بهم:

في حالة وجود أسئلة محدّدة تتعلّق بهذا البحث ، أو في حالة حدوث أي إصابات تتصل بالدراسة ناتجة عن المشاركة بالدراسة ، نرجو الاتصال على الباحث الرئيسي/نانبه. دكتورة / جينيفر دي بير هاتف رقم ۱۲۲۲۷۷۷۷۰- تحویلة رقم ... 66403 للأسئلة العامة المتعلقة بالبحوث بمستشفى الملك فيصل التخمتصي ومركز الأبحاث بجدة يرجى الإتصال على منسقة الأبحاث على هاتف رقم ١٢٦٦٧٧٧٧٧ تحويلة رقم 63537. أو الاتصال على رئيس لجنة أخلاقيات الأبحاث /نائبه ......على هاتف رقم

ل. إقرار الباحث الرئيس إنانبه:

.966114424528

#### L. I, the principal investigator/delegate

I Dr / Jennifer de Beer have fully explained to the above (volunteer/ guardian)\* the nature and purpose of the above-mentioned research program (including the fact that the studies will not result in any direct therapeutic benefit and the extent, if any, to which the studies are experimental), the possible complications اقر أنا دكتورة / جينيفر دي بير

بانني قد شرحت (المتطوع/ أو ولي امره الشرعي) \* المذكور اعلاه بصورة كاملة طبيعة وأهداف مشروع البحث المذكور والمتضمن عدم وجود فاندة مباشرة على المشارك\* والي أي مدى (إن وجد) هي دراسة تجريبية, كما قد شرحت المضاعفات المحتمل حدوثها من جراء هذه الدراسة سواء كانت لأسباب معروفة أو غير معروفة والعواقب والمخاطر المترتبة (إن وجدت) إذا قرر المتطوع إنهاء مشاركته بالدراسة.

This Informed Consent Form (ICF) is approved by the KFSHRC -IRB

IRB # 2251201

Approval Dated:

ICF Version No.: 1.0

From: 27 October 2025

To: 31 August 2026



which may arise from both known and unknown causes as a result thereof and the consequences and risks, if any, if the volunteer decides to discontinue participation.

It is my understanding that he/she understands the nature, purposes, and risks of these studies before he signs this informed consent. I have also offered to answer any questions relating to these studies and have fully and completely answered all such questions.

كما إنه من المفهوم لدي بأنه قد فهم طبيعة الدراسة والغرض منها والمخاطر الناتجة عنها وذلك قبل توقيعه على الموافقة بالمشاركة ، ولقد قمت بتوضيح استعدادي للإجابة على أي أسئلة متصلة بهذه الدراسة ، وقمت فعلاً بالإجابة الشافية على جميع أسئلته المتعلقة بالدراسة.

This Informed Consent Form (ICF) is approved by the KFSHRC -IRB

ICF Version No.: 1.0

IRB # 2251201

Approval Dated:

From: 27 October 2025

To: 31 August 2026 🍱



### PART II: Authorization of Voluntary participant:

# الجزء الثاني: تفويض من المشارك بالدراسة:

M. I, the the participate acknowledge that I have read (or it had been explained to me in a clear language) the attached Research Participant Information Form and Dr/ Jennifer de Beer

has explained to me the nature and purpose of this study in this form, as well as any reasonably expected benefits, possible alternative methods of treatment, the attendant discomforts and risks reasonably expected, and the possibility that complications from both known and unknown causes may arise as a result thereof. I have had the opportunity to ask any questions I had regarding this study and all those questions were answered to my satisfaction.

م. أقر أنا المشارك بأنني قد قرأت (أو قد شرحت لي بلغة واضحة) جميع المعلومات الموجودة في نموذج الإقرار بالموافقة على المشاركة بالأبحاث وإن دكتورة / جينيفر دي بير قد أوضح لي ماهية الدراسة في هذا النموذج والغرض منها والفوائد المرجوة منها والطرق العلاجية البديلة لها, والمخاطر أوالانز عاجات المتوقع حدوثها, وكذلك احتمال حدوث مضاعفات السباب معروفة أو غير معروفة نتيجة لذلك. كما أنه قد أتيحت لى الفرصة الكافية لطرح أي سؤال يتعلِّق بالدراسة وتلقيت الإجابات الكافية

I acknowledge I do not have any preexisting medical or emotional problem which would make it unwise for me to participate in these studies.

كما أقر بأنني لا أعاني من أي مشاكل طبية أو نفسية معروفة لدى بحيث قد يكون من غير الحكمة أن أشارك بهذه الدراسة.

Based on the above mentioned information I voluntarily accept participation in this research study and I understand that I am free to withdraw this consent and discontinue my participation in this study at any time. The consequences and risks, if any, which might be involved if I decided to discontinue my participation have been explained to me. I understand that such withdrawal will not affect my ability to receive any medical care to which I might be otherwise entitled.

بناء على ما سبق و بمحض إر ادتى فإني أنطوع بالمشاركة في هذه الدر اسة. وافهم أن لي مطلق الحرية بسحب موافقتي وقطع مشاركتي بالدراسة في أي وقت. هذا وقد شرحت لي جميع العواقب والمخاطر المترتبة (إن وجدت) عن انسحابي من الدر اسة. كما أفهم بأن انسحابي من هذه الدر اسة لن يؤثر في حقى في تلقّى العناية الطبية اللازمة التي استحقها في الأحوال العادية.

This Informed Consent Form (ICF) is approved by the KFSHRC -IRB

ICF Version No.: 1.0

IRB # 2251201

Approval Dated:

From: 27 October 2025

To: 31 August 2026 🍱



| Title of Research: A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses | عنوان البحث: تجربة سريرية عشوانية مضبوطة حول تطبيق الذكاء<br>الاصطناعي في تقييم الجلد للوقاية من تقرحات الفراش وتحديد مراحلها<br>بواسطة ممرضي وحدات العناية المركزة |
|---|---|
| Name of Participant: | اسم المشارك: |
| Name of individual signing the consent form: | اسم الموقع على هذا الإقرار: |
| Gaurdian's Relation*: | صفة ولي الأمر*: |
| Signature: | التوقيع: |
| Date: | التاريخ: |
| I confirm that I have accurately (translated and/ or read)* the information to the subject: | اقر بانني قد (قرأت / أو ترجمت) * للمشارك هذه المعلومات بدقة<br>اسم الشاهد : |
| Witness Name: | |
| Signature/(National I.D./Iqama/Hospital I.D. No.): | التوقيع/ (رقم الهوية/ الإقامة/ الرقم الوظيفي): |
| Date / Time: | التاريخ/ الوقت: |
| Signature of Principal Investigator/ Delegate | توقيع الباحث الرنيسي/نانيه |
| Name: Dr Jennifer de Beer | الأسم: |
| I.D. No.: 69129 | الرقم الوظيفي: |
| Title:Nursing Research Senior Specialist | الوظيفة: |
| Signature: | التوقيع: |
| Date: | التاريخ: |

This Informed Consent Form (ICF) is approved by the KFSHRC -IRB

ICF Version No.: 1.0

IRB # 2251201

Approval Dated:

From: 27 October 2025

To: 31 August 2026 🏝

